CLINICAL TRIAL: NCT04906616
Title: An Economic and Relationship-strengthening Intervention for HIV-affected Couples Who Drink Alcohol in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Invest in Knowledge Initiative (IKI) - Zomba, Malawi (Other); University of Michigan (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P0535590; R34AA027983-01 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: HIV/AIDS; Alcohol Abuse
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcoholism

STUDY DESIGN:
Intervention Model Description: Couples will be randomized 1:1 to intervention or control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Comparison (No Intervention): Standard of care, e.g. regular HIV care plus brief advice on alcohol use
- Mlambe Intervention (Experimental): A couples-based intervention to reduce problematic drinking and improve economic and HIV outcomes.
  Interventions: Behavioral: Mlambe

INTERVENTIONS:
Behavioral: Mlambe — A combined economic and relationship-strengthening intervention at the couple level to redirect funds spent on alcohol into financial investments (e.g., education, income-generating business) and to improve couple relationships and adherence to ART.
  Arms: Mlambe Intervention

SUMMARY:
A couples-based alcohol-reduction and economic and relationship-strengthening intervention for HIV-affected couples in Malawi.

DETAILED DESCRIPTION:
This project aims to develop and pilot test a combined economic and relationship-strengthening intervention to redirect funds spent on alcohol into financial investments (e.g., education, income-generating business) and to improve couple relationships and adherence to ART. The study hypothesizes that engaging couples to work together on alcohol use and financial goals-equipped with financial, communication, and problem-solving skills-will decrease alcohol use, and improve relationship dynamics and adherence to ART. Specifically, the project aims: (1) to adapt and integrate two proven interventions, Suubi and Uthando Lwethu, using the ADAPT-ITT method, into a combined intervention for HIV-affected couples with a heavy alcohol user (to be called Mlambe); (2) to develop and pilot test the study procedures to evaluate Mlambe; and (3) to assess the feasibility and acceptability of Mlambe through a pilot study. In the formative phase, the study will develop a draft of the intervention manual and conduct five focus group discussions with couples and key stakeholders to obtain input on the intervention. In the pilot phase, 80 HIV-affected couples with a heavy alcohol user will be enrolled and randomized to either Mlambe or the comparison arm (regular HIV care plus brief advice on alcohol use). The study will conduct qualitative interviews with a subset of 20 couples to contextualize feasibility and acceptability data, and then will analyze the mixed- methods feasibility and acceptability data to refine intervention and procedures for a future trial.

ELIGIBILITY:
Inclusion Criteria:

* in a married or cohabitating union
* have at least one partner with a positive AUDIT-C screen in prior 3 months who is also currently on ART for at least 6 months who has disclosed their HIV status to their partner

Exclusion Criteria:

* severe intimate partner violence reported in previous 3 months and/or fear that safety would be at risk by participation in the study (reported at screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Conroy, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Invest in Knowledge Initiative (IKI), Zomba, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conroy A, Leddy A, Johnson M, Ngubane T, van Rooyen H, Darbes L. 'I told her this is your life': relationship dynamics, partner support and adherence to antiretroviral therapy among South African couples. Cult Health Sex. 2017 Nov;19(11):1239-1253. doi: 10.1080/13691058.2017.1309460. Epub 2017 Apr 11. PMID 28398134
- [Background] Conroy AA, McKenna SA, Ruark A. Couple Interdependence Impacts Alcohol Use and Adherence to Antiretroviral Therapy in Malawi. AIDS Behav. 2019 Jan;23(1):201-210. doi: 10.1007/s10461-018-2275-2. PMID 30218319
- [Background] Conroy AA, Ruark A, McKenna SA, Tan JY, Darbes LA, Hahn JA, Mkandawire J. The Unaddressed Needs of Alcohol-Using Couples on Antiretroviral Therapy in Malawi: Formative Research on Multilevel Interventions. AIDS Behav. 2020 Jun;24(6):1599-1611. doi: 10.1007/s10461-019-02653-y. PMID 31456201
- [Background] Darbes LA, McGrath NM, Hosegood V, Johnson MO, Fritz K, Ngubane T, van Rooyen H. Results of a Couples-Based Randomized Controlled Trial Aimed to Increase Testing for HIV. J Acquir Immune Defic Syndr. 2019 Apr 1;80(4):404-413. doi: 10.1097/QAI.0000000000001948. PMID 30730356
- [Background] Ssewamala FM, Han CK, Neilands TB. Asset ownership and health and mental health functioning among AIDS-orphaned adolescents: findings from a randomized clinical trial in rural Uganda. Soc Sci Med. 2009 Jul;69(2):191-8. doi: 10.1016/j.socscimed.2009.05.019. Epub 2009 Jun 10. PMID 19520472
- [Background] Bermudez LG, Ssewamala FM, Neilands TB, Lu L, Jennings L, Nakigozi G, Mellins CA, McKay M, Mukasa M. Does Economic Strengthening Improve Viral Suppression Among Adolescents Living with HIV? Results From a Cluster Randomized Trial in Uganda. AIDS Behav. 2018 Nov;22(11):3763-3772. doi: 10.1007/s10461-018-2173-7. PMID 29846836
- [Derived] Gopalakrishnan L, Mulauzi N, Mkandawire J, Ssewamala FM, Tebbetts S, Neilands TB, Conroy AA. Effects of economic empowerment and relationship strengthening intervention on financial behaviors among couples living with HIV: The Mlambe pilot trial in Malawi. SSM Popul Health. 2025 Feb 25;29:101768. doi: 10.1016/j.ssmph.2025.101768. eCollection 2025 Mar. PMID 40104040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The values in the data table represent individual participants and not couples.
Period: Overall Study
Arm/Group | Control Comparison | Mlambe Intervention
Started | 78 | 78
Completed | 75 | 76
Not Completed | 3 | 2
Not completed — Divorce | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Comparison | Mlambe Intervention | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (10.3) | 43.2 (10.1) | 43.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 39 | 39 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 78 | 78 | 156
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 78 | 78 | 156

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Percentage of eligible couples enrolled in the study.
Time Frame: Baseline (Time 0)
Population: 89 couples were screened as eligible for inclusion in the study. 84 couples completed baseline assessments. 78 couples (156 participants) were randomized into the study: 39 couples into the control arm and 39 couples into the intervention arm.
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Groups:
- Enrollment Rate: Percentage of eligible couples who completed baseline assessments.
Arm/Group | Enrollment Rate
Number analyzed (Participants) | 178
Number analyzed (couples) | 89
couples | 84

2. Primary Outcome: Retention Rate
Description: Percentage of enrolled and randomized participants retained at the end of the study
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Participants | 75 | 76

3. Secondary Outcome: Percentage of Couples Who Are "Satisfied" or "Very Satisfied" With the Intervention at 10 Months
Description: Percentage of couples reporting to be "satisfied" or "very satisfied" about their overall experience with the Mlambe intervention on a five-point scale (the Mlambe Satisfaction Survey) at 10 months. Response options included: (1) very satisfied; (2) satisfied; (3) neutral; (4) unsatisfied; (5) very unsatisfied.
Time Frame: 10 months
Population: This count here is for couples, not individuals.
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Number analyzed (couples) | 39 | 39
couples | 39 | 39

4. Secondary Outcome: Percentage of Couples Who Are Satisfied With the Intervention at 15 Months
Description: Percentage of couples reporting to be "satisfied" or "very satisfied" about their overall experience with the Mlambe intervention on a five-point scale (the Mlambe Satisfaction Survey) at 15 months. Response options included: (1) very satisfied; (2) satisfied; (3) neutral; (4) unsatisfied; (5) very unsatisfied.
Time Frame: 15 months
Population: The units analyzed are for couples (not individuals)
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Number analyzed (couples) | 39 | 39
couples | 39 | 39

5. Secondary Outcome: 10 Month Follow up Survey Completion
Description: Percentage of couples who complete follow up surveys at 10 months
Time Frame: 10 months
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Number analyzed (couples) | 39 | 39
couples | 36 | 38

6. Secondary Outcome: 15 Month Follow up Survey Completion
Description: Percentage of couples who complete follow up surveys at 15 months
Time Frame: 15 months
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Number analyzed (couples) | 39 | 39
couples | 37 | 37

7. Secondary Outcome: 75% Intervention Completion
Description: Percentage of couples who attend 75% of intervention sessions
Time Frame: 10 months
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Number analyzed (couples) | 39 | 39
couples | 39 | 39

8. Secondary Outcome: 100% Intervention Completion
Description: Percentage of couples who attend 100% of intervention sessions
Time Frame: 10 months
Measure: Count of Units; unit: couples
Units Other Than Participants: couples
Arm/Group | Control Comparison | Mlambe Intervention
Number analyzed (Participants) | 78 | 78
Number analyzed (couples) | 39 | 39
couples | 39 | 39

9. Other Pre Specified Outcome: Exploratory: Alcohol Use
Description: Number of drinking days in the past 21 days, assessed via the Timeline Follow-Back Method
Time Frame: 10 months, 15 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory: Alcohol Use
Description: Non-heavy drinking determined by self-report (Alcohol Use Disorders Identification Test - Consumption [AUDIT-C], prior 3 months, negative) and phosphatidylethanol (PEth) <35 ng/mL (composite measure)
Time Frame: 10 months, 15 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory: Viral Suppression
Description: Proportion of HIV-infected participants who are virally suppressed by local lab normal ranges, as measured by dried blood spots (DBS)
Time Frame: 10 months, 15 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory: ART Adherence
Description: Proportion of pills taken by HIV-infected participants in the past 30 days, using the bean count method (self-report) adapted from VAS
Time Frame: 10 months, 15 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Control Comparison | Mlambe Intervention
All-Cause Mortality (participants affected / at risk) | 0/78 | 1/78
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 0/78 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT04906616/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT04906616/ICF_001.pdf